CLINICAL TRIAL: NCT06625372
Title: Comparison of the Effect of Intralipid Parenteral Nutritional With SMOF Lipid Parenteral Nutritional on Biochemical Markers, Hematologic Markers, and Clinical Outcomes Following Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Comparison of Intralipid With SMOF Lipid Following HSCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Associate professor, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 0311.212
Record Dates: First submitted 2024-09-28; First posted 2024-10-03 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Leukemia; HSCT
Keywords: mortality; SMOF; Intralipid; Engrafment; Complications
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMOF lipid (Experimental): The SMOF lipid is given to the patient as a fat component of total parenteral nutrition.
  Interventions: Dietary Supplement: SMOF lipid
- Intralipid (Active Comparator): intralipids
  Interventions: Dietary Supplement: INTRALIPIDS

INTERVENTIONS:
Dietary Supplement: SMOF lipid — The SMOF lipid is given to the patient as a fat component of total parenteral nutrition.
  Arms: SMOF lipid
Dietary Supplement: INTRALIPIDS — The Intralipid will be given to the patient as fat component of total parenteral nutrition.
  Arms: Intralipid

SUMMARY:
The goal of this clinical trial is to have a successful engraftment in after bone transplantation. Acute leukemia patient of both sexes aged 2 to 18 years, who are transplant candidates, participate in this study. Primary hypothesis is Patients receiving SMOF LIPID will have better grafts than patients receiving intralipid. Also, complications after surgery and malnutrition will be less in this group.

DETAILED DESCRIPTION:
Patients will be randomly divided into two groups: the intervention group (TPN based on SMOFLipid) and the control group (TPN based on IntraLipid). At baseline (before HSCT) and after obtaining informed consent and assent, blood samples will be collected to test for biochemical markers, including total cholesterol, TG, LDL, HDL, FBS, Alb, Na, K, Ph, Ca, Mg, CRP, IL-6, BUN, Cr, and CBC. Furthermore, data on nutritional intake (total energy and protein) and appetite status will be gathered. The primary outcomes are neutrophil and platelet engraftment, defined as >500 for neutrophils and >20,000 for platelets, respectively. The possibility of oral intake, as well as the achievement of oral + ONS and total oral nutrition alongside TPN duration, will be recorded. On days +15 and +30, biochemical and anthropometric markers will be collected again. Furthermore, clinical outcomes such as acute GVHD, cholestasis, bleeding, infections, hospitalization, and mortality will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to cooperate and complete the informed consent form by the legal guardian of the child;
* Age ≤ 18 years;
* Definitive diagnosis of acute leukemia and candidate for hematopoietic stem ● cell transplantation;
* Eligible for parenteral nutrition support;
* No contraindications for parenteral nutrition;
* No history of allergy to egg or soy protein;
* Absence of severe organ failure or impaired liver function test (bilirubin > 2.5 mg/dL).

Exclusion Criteria:

* Death of the child earlier than 5 days from the start of the intervention;
* Unwillingness to continue cooperation during study;
* Occurrence of side effects during the study;
* In case of sepsis, hypotension, shock, thrombosis, myocardial infarction, liver dysfunction, the patient will be excluded from the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Engraftment | Within 35 days after transplantation
  blood counts of Neutrophils and platelets

SECONDARY OUTCOMES:
100-day survival rate | Within 100 days after transplantation
  Determination and comparison of 100-day survival rate after transplantation in both groups
Incidence of infection | Within 30 days after transplant
  Determining and comparing the incidence of infection
Incidence of bleeding | Within 30 days after transplantation
  Determining and comparing the incidence of bleeding
Hospitalization | up to 7 weeks after transplantation
  Determining and comparing the duration of hospitalization in both groups
Mortality | up to 7 weeks after transplantation
  incidence of mortality in hospital
MAC (mid arm circumference) | On days 15 and 30 after transplantation
  Determination and comparison of MAC in both groups
Albumin | On days 15 and 30 after transplantation
  Determination and comparison of serum albumin
Acute gastrointestinal complications | Up to 100 days after transplantation
  Determining and comparing the incidence of acute gastrointestinal complications (including acute GVHD, cholestasis) in both groups.
Duration of parenteral nutrition | during hospitalization, up to 7 weeks after transplantation
  Determining and comparing the duration of using parenteral nutrition
Weight | On days 15 and 30 after transplantation
  Determination and comparison of weight in both groups
Blood sugar | On days 15 and 30 after transplantation
  Determination and comparison of blood sugar,
Serum electrolytes | On days 15 and 30 after transplantation
  Determination and comparison of serum electrolytes
Serum lipids | On days 15 and 30 after transplantation
  Determination and comparison of serum lipids
Serum Interleukin 6 (IL-6) | On days 15 and 30 after transplantation
  Determination of serum interleukin 6 (IL-6)

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Vahdat Shariatpanahi, Professor, Principal Investigator — School of Nutrition Sciences and Food Technology, Shahid Beheshti University of Medical Sciences
Locations (1):
- Children's Medical Center, Pediatrics Center of Excellence, Tehran University of Medical Sciences, Tehran, Iran, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No